CLINICAL TRIAL: NCT01134887
Title: Controlling Hypertension Outcomes by Improved Communication & Engagement (CHOICE)
Brief Title: Controlling Hypertension Outcomes by Improved Communication & Engagement
Acronym: CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RRP 09-190
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-06

CONDITIONS: Hypertension; Stroke
Keywords: hypertension; physician-patient relations; communication
MeSH Terms: conditions — Hypertension; Stroke; Communication | interventions — Physicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Intervention-Veterans (Experimental): Veterans enrolled in the "Intervention-Veterans" arm received a copy of the NIA guide for "Talking with Your Doctor" [Informational Guide for Patients]. Just prior to their next scheduled visit an educator met with each Veteran in the intervention arm individually for 20-30 minutes to review the material in the pamphlet and develop a plan for enhancing communication about self-management of hypertension with their doctor [Educational Coaching]. To facilitate communication change, the educator assisted the patient in setting a goal to achieve during their visit. The educator also provided telephone follow-up within 24 hours to review satisfaction and effectiveness of the visit and assess barriers and facilitators to communicating about self-management.
  Interventions: Other: Informational Guide for Patients; Behavioral: Educational Coaching
- Arm 2: Control-Veterans (Active Comparator): Veterans enrolled in the "Control-Veterans" arm received a copy of the NIA guide for "Talking with Your Doctor" [Informational Guide for Patients]. This pamphlet was specifically developed for this purpose (updated in 2002). It has pictorials and is written at an 8th grade level.
  Interventions: Other: Informational Guide for Patients
- Arm 3: Intervention-Physicians (Experimental): Primary care providers randomly assigned to the "Intervention-Physicians" arm of this study received a copy of the Four Habits of Highly Effective Physicians [Monograph for Physicians]. The Four Habits provided practical evidence-based advice for improving patient-physician communication. Second, physicians participated in an audiotaped intensive 30 minute, one-on-one educational intervention with PI Frankel after their first set of visits from their three participating patients [Video-Assisted Coaching], but before seeing them for follow-ups. The main goal of this meeting was to review and discuss the analysis of the physician's videotaped visits using the Four Habits framework, with a particular focus on improving communication about self-management.
  Interventions: Behavioral: Video-Assisted Coaching; Other: Monograph for Physicians
- Arm 4: Control-Physicians (Active Comparator): Primary care providers randomly assigned to the "Control-Physicians" arm of the study did not receive coaching or additional resources, and conducted their primary care practice as usual [Control].
  Interventions: Other: Control

INTERVENTIONS:
Other: Informational Guide for Patients — Veterans received a copy of the NIA guide for "Talking with Your Doctor". This pamphlet was specifically developed for this purpose (updated in 2002). It has pictorials and is written at an 8th grade level.
  Arms: Arm 1: Intervention-Veterans; Arm 2: Control-Veterans
Behavioral: Video-Assisted Coaching — Physicians participated in an audiotaped intensive 30 minute, one-on-one educational intervention with PI Frankel after their first set of visits from their three participating patients, but before seeing them for follow-ups. The main goal of this video-assisted coaching session was to review and discuss the analysis of the physician's videotaped visits using the Four Habits framework, with a particular focus on improving communication about self-management.
  Arms: Arm 3: Intervention-Physicians
Other: Monograph for Physicians — Primary care providers randomly assigned to the "Intervention-Physicians" arm of this study received a copy of the Four Habits of Highly Effective Physicians. The Four Habits provided practical evidence-based advice for improving patient-physician communication.
  Arms: Arm 3: Intervention-Physicians
Behavioral: Educational Coaching — an educator met with each Veteran in the intervention arm individually for 20-30 minutes to review the material in the pamphlet and develop a plan for enhancing communication about self-management of hypertension with their doctor [Coaching]. To facilitate communication change, the educator assisted the patient in setting a goal to achieve during their visit. The educator also provided telephone follow-up within 24 hours to review satisfaction and effectiveness of the visit and assess barriers and facilitators to communicating about self-management.
  Arms: Arm 1: Intervention-Veterans
Other: Control — The primary care providers randomly assigned to the "Control-Physicians" arm did not receive any additional coaching or resources and conducted their practice as usual.
  Arms: Arm 4: Control-Physicians

SUMMARY:
This randomized control study tested the feasibility of two communication enhancement interventions: one with veterans who had a stroke and demonstrated poorly controlled hypertension; the other with VA primary care providers who provided routine outpatient medical care to these veterans. This study intervened with both members of the provider-patient dyad in an attempt to improve the self-management of hypertension by improving communication during visits to the VA outpatient clinic, specifically by enabling veterans to communicate their questions and concerns about chronic disease self-management to their providers more effectively, and to help providers improve their ability to communicate more effectively with this population of veterans.

DETAILED DESCRIPTION:
The communication intervention had two goals; (a) coaching to enhance veteran's abilities to communicate their questions and concerns about self-management for hypertension to their physician; and (b) improving provider's communication skills for enhancing and encouraging self-management of hypertension.

A health educator met with each participating veteran in the intervention arm prior to the 2nd visit to develop a plan for enhancing communication about self-management of hypertension.

The PI provided the Four Habits communication training to the 5 primary care providers in the intervention arm. Two clinic visits between each participating provider-patient pair were videotaped and coded.

This project had a goal of enrolling 10 VA primary care providers to participate in the randomized control trial and 30 veterans (3 veterans from the panel of each of the 10 participating providers) who had a stroke and now demonstrated poorly controlled hypertension. The study evaluated the difference between the two groups, and compared the content of the provider-patient conversations around hypertension management.

ELIGIBILITY:
Inclusion Criteria:

Veteran:

* Veteran is a patient of the enrolled provider
* History of prior stroke
* Poorly controlled hypertension with at least one measurement >140/90 mm Hg in the past 12 months
* Complete a 6-item screen for cognitive and language impairment with a score of 3 or higher
* Sign the VA Media consent for use of picture and/or voice

Provider:

* Primary care provider, Medicine Service
* Sign VA media consent for use of picture and/or voice

Exclusion Criteria:

* Life expectancy is less than 6 months
* Non-English language patients
* Inability to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2012-09-30 (Actual); Study Completion 2017-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Frankel, PhD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (2):
- United States (2):
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten physicians and 20 Veterans were recruited into the study at the Roudebush VA Medical Center in Indianapolis, Indiana. The 20 Veterans were patients in the panels of the ten participating physicians. Four patients did not complete the protocol reducing the overall number of completers to 26.
Groups:
- Arm 1: Intervention-Veteran: Veterans enrolled in the "Intervention-Veterans" arm received a copy of the NIA guide for "Talking with Your Doctor." Just prior to their next scheduled visit an educator met with each Veteran in the intervention arm individually for 20-30 minutes to review the material in the pamphlet and develop a plan for enhancing communication about self-management of hypertension with their doctor. To facilitate communication change, the educator assisted the patient in setting a goal to achieve during their visit. The educator also provided telephone follow-up within 24 hours to review satisfaction and effectiveness of the visit and assess barriers and facilitators to communicating about self-management.
- Arm 2: Control-Veteran: Veterans enrolled in the "Control-Veterans" arm received a copy of the NIA guide for "Talking with Your Doctor." This pamphlet was specifically developed for this purpose (updated in 2002). It has pictorials and is written at an 8th grade level.
- Arm 3: Intervention-Physician: Primary care providers randomly assigned to the "Intervention-Physicians" arm of this study received a copy of the Four Habits of Highly Effective Physicians. The Four Habits provided practical evidence-based advice for improving patient-physician communication. Second, physicians participated in an audiotaped intensive 30 minute, one-on-one educational intervention with PI Frankel after their first set of visits from their three participating patients, but before seeing them for follow-ups. The main goal of this meeting was to review and discuss the analysis of the physician's videotaped visits using the Four Habits framework, with a particular focus on improving communication about self-management.
- Arm 4: Control-Physician: Primary care providers randomly assigned to the "Control-Physicians" arm of the study did not receive coaching or additional resources, and conducted their primary care practice as usual.
Period: Overall Study
Arm/Group | Arm 1: Intervention-Veteran | Arm 2: Control-Veteran | Arm 3: Intervention-Physician | Arm 4: Control-Physician
Started | 9 | 11 | 5 | 5
Completed | 9 | 7 (Four patients in the Veteran-Control arm did not have two clinic visits videotaped and left study.) | 5 | 5
Not Completed | 0 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Intervention-Veteran | Arm 2: Control-Veteran | Arm 3: Intervention-Physician | Arm 4: Control-Physician | Total
Number analyzed (Participants) | 9 | 11 | 5 | 5 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 5 | 5 | 21
  >=65 years | 4 | 5 | 0 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 3 | 4 | 7
  Male | 9 | 11 | 2 | 1 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 11 | 5 | 5 | 30
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 5 | 5 | 30

OUTCOME MEASURES:

1. Primary Outcome: Patient Activation Measure
Description: Veteran self-management of hypertension measured via the 13-item, (0-100 point range), Patient Activation Measure (PAM). Administered at baseline (1st visit) and after each additional follow-up visit during the next 12-months (+2 max). Rasch conversion changed raw scores to the PAM interval measure. Reported outcome is difference in mean PAM scores at baseline and during 12-month follow-up. If a participant had two PAM scores during the follow-up period, the average of the two was taken to calculate a combined follow-up score. Higher PAM scores represent higher levels of self-activation. Research on the PAM measure indicates that each point increase in PAM score correlates to a 2% decrease in hospitalization and a 2% increase in medication adherence. Ranges for Baseline PAM scores: Intervention = 46.1 (min) to 84.3 (max); Control = 43.2 (min) to 77 (max). Ranges for Follow-up PAM scores: Intervention = 48.4 (min) to 100 (max); Control = 45.1 (min) to 80.1 (max).
Time Frame: 12 months
Population: Veterans participating in CHOICE study randomized to two arms: intervention or attention control. The 13-item Patient Activation Measure was administered at baseline and up to two additional times during the following 12 months. Rasch conversion of the raw PAM scores was performed to ensure the final scores were linear and interval measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Intervention-Veterans: Veterans randomized to the intervention group received a copy of the NIA guide for "Talking with Your Doctor." Just prior to their next scheduled visit, an educator met with each Veteran in the intervention arm individually for 20-30 minutes to review the material in the pamphlet and develop a plan for enhancing communication about self-management of hypertension with their doctor. Additional information was provided on how to be an active participant in the health care encounter and how to communicate effectively to promote productive self-management. To facilitate communication change, the educator assisted the Veteran in setting a goal to achieve during their visit. The educator also provided telephone follow-up within 24 hours to review satisfaction and effectiveness of the visit and assess barriers and facilitators to communicating about self-management.
- Arm 2: Control-Veterans: The attention control comparator consisted of giving Veterans a copy of the NIA guide for "Talking with Your Doctor." This pamphlet was specifically developed for this purpose (updated in 2002). It has pictorials and is written at an 8th grade level.
Arm/Group | Arm 1: Intervention-Veterans | Arm 2: Control-Veterans
Number analyzed (Participants) | 9 | 11
units on a scale
  Baseline PAM | 61.33 (13.39) | 60.86 (11.41)
  Followup PAM | 63.49 (14.45) | 57.45 (8.65)

ADVERSE EVENTS:
Groups:
- Arm 1: Intervention: Veterans enrolled in the intervention arm received a copy of the NIA guide for "Talking with Your Doctor." Just prior to their next scheduled visit an educator met with each Veteran in the intervention arm individually for 20-30 minutes to review the material in the pamphlet and develop a plan for enhancing communication about self-management of hypertension with their doctor. Additional information was provided on how to be an active participant in the health care encounter and how to communicate effectively to promote productive self-management. To facilitate communication change, the educator assisted the patient in setting a goal to achieve during their visit. The educator also provided telephone follow-up within 24 hours to review satisfaction and effectiveness of the visit and assess barriers and facilitators to communicating about self-management.
- Arm 2: Attention Control: Veterans enrolled in the attention control arm received a copy of the NIA guide for "Talking with Your Doctor." This pamphlet was specifically developed for this purpose (updated in 2002). It has pictorials and is written at an 8th grade level.
- Arm 3: Intervention-Physicians: The 5 intervention arm physicians were coached in the Four Habits of Highly Effective Clinicians in a one hour face to face meeting involving review of the provider's interaction with his or her intervention patients and suggestions for improvement based on these observations.
- Arm 4: Control-Physicians: Control physicians were told to conduct their encounters as usual and were not given any coaching. Adverse event reporting was provided as part of the study.
Arm/Group | Arm 1: Intervention | Arm 2: Attention Control | Arm 3: Intervention-Physicians | Arm 4: Control-Physicians
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes